CLINICAL TRIAL: NCT05691933
Title: Ultrasound Guided External Oblique Intercostal Plane Block for Perioperative Analgesia in Major Upper Abdominal Surgery: Prospective Randomized Controlled Study
Brief Title: Regional Block for Upper Abdominal Surgeries
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0305400
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Perioperative Analgesia in Major Upper Abdominal Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block group (Active Comparator): Patients will be subjected to bilateral external oblique intercostal plane block
  Interventions: Procedure: Block group
- Opioid group (Active Comparator): Patients will be subjected to morphine infusion at a rate of 0.03mg/kg/h
  Interventions: Procedure: Morphine infusion

INTERVENTIONS:
Procedure: Block group — Patient will be subjected to bilateral external oblique intercostal plane block
  Arms: Block group
Procedure: Morphine infusion — Patients will be subjected to morphine infusion at a rate of 0.03mg/kg/h
  Arms: Opioid group

SUMMARY:
Pain control after major upper abdominal surgeries is an essential step to guard against postoperative complications such as lung atelectasis. This major step can be achieved by opioids or regional blocks.

Regional blocks allow better pain control and avoid side effects of opioid based pain control

DETAILED DESCRIPTION:
Ultrasound guided External oblique intercostal plane block for perioperative analgesia in major upper abdominal surgery: Prospective randomized controlled study

Introduction:

Pain control is a vital component to achieve enhanced recovery after major upper abdominal surgery. Effective postoperative pain control will reduce the incidence of numerous postoperative complications, can facilitate early mobilization and may result in earlier recovery.

Pain control is historically achieved by the administration of opioids, which is associated with well-documented side effects, such as sedation, respiratory depression, pruritus, hallucinations and postoperative nausea and vomiting (PONV). Epidural analgesia, another routinely used analgesic technique, offers equivalent or superior pain scores when compared to conventional systemic opioids. Enhanced recovery following major upper abdominal surgery has gained attention even though there is limited evidence on the efficacy and effectiveness of existing analgesic techniques.

The external oblique intercostal plane block is a new modality that will be used to improve pain-related outcomes after major upper abdominal surgeries, and has not been extensively investigated. Therefore, we will test the hypothesis that external oblique intercostal plane block can reduce cumulative opioid consumption for the patients undergoing major upper abdominal surgery when added to conventional multi-model intravenous analgesic technique.

The aim of this prospective comparative investigation is to assess the impact of external oblique intercostal plane block in a multimodal perioperative analgesic regimen and any related side effects in patients undergoing major upper abdominal surgery.

Patients and Methods:

A prospective study will be carried out in Alexandria Main University Hospital on 120 American society of anaesthesiologists (ASA) II, III physical status aged 20-60 years scheduled for major upper abdominal surgery, after approval of the Medical Ethics Committee and an informed written consent. Patients will be categorized into two equal groups, group I (60) will be subjected to bilateral external oblique intercostal plane block and group II (60) will be subjected to morphine infusion at a rate of 0.03mg/kg/h. During the patient stay in the ICU, total analgesic requirements will be measured in both groups. Also, sedation level, duration of intubation and length of ICU stay will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing upper abdominal surgeries

Exclusion Criteria:

* BMI above 40

  * allergy for drugs used
  * complicated cases
  * patient refusal
  * chronic opioid use
  * cognitive dysfunction
  * chronic kidney disease
* Liver failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative morphine requirements for 24 hours | 24 hours postoperatively
  Visual analogue score will be measured every 2 hours

SECONDARY OUTCOMES:
Pain assessment | 24 hours postoperatively
  Visual analogue score will be assessed every 2hours postoperatively
Rescue analgesia | 24 hours postoperatively
  0.5 microgram/kg fentanyl will be given if VAS score more than 4
Side effects | 24 hours postoperatively
  Any side effect related to fentanyl or block

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on request
Supporting Information: Study Protocol, ICF
Time Frame: One year
URL: http://www.alexu.edu.eg

REFERENCES:
- [Background] Hughes M, McNally S, McKeown DW, Wigmore S. Effect of analgesic modality on outcome following open liver surgery: a systematic review of postoperative analgesia. Minerva Anestesiol. 2015 May;81(5):541-56. Epub 2014 Jun 11. PMID 24918191
- [Background] Rosero EB, Cheng GS, Khatri KP, Joshi GP. Evaluation of epidural analgesia for open major liver resection surgery from a US inpatient sample. Proc (Bayl Univ Med Cent). 2014 Oct;27(4):305-12. doi: 10.1080/08998280.2014.11929141. PMID 25484494